CLINICAL TRIAL: NCT00153517
Title: Maternal Effects of Bacterial Vaginosis (BV) Treatment in Pregnancy (Randomized Trial of BV Treatment in Pregnancy)
Brief Title: Maternal Effects of Bacterial Vaginosis (BV) Treatment in Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cynthia Ferre, Lead Health Scientist, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDC-NCCDPHP-2752; U36CCU300430-2239 (Other Grant/Funding Number: CDC); U36CCU300430-1179 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Vaginosis, Bacterial; Premature Birth; Birth Weight; Chorioamnionitis
Keywords: Bacterial Vaginosis; Metronidazole
MeSH Terms: conditions — Vaginosis, Bacterial; Premature Birth; Birth Weight; Chorioamnionitis

STUDY DESIGN:
Intervention Model Description: study participants were randomized to treatment with oral metronidazole (Centers for Disease Control and Prevention [CDC] recommended regimen: 250mg three times daily for 7 days) plus intravaginal placebo or intravaginal metronidazole (5 g of 0.75% gel twice daily for 5 days) plus oral placebo. The oral and vaginal placebos were indistinguishable from active therapy. Randomization to study group used random number tables, with a 1:1 ratio between study groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Investigational Drug Service at the University of Washington performed the randomization and provided the treatment assignments in opaque, sealed envelopes. Neither the subjects nor the study personnel assessing treatment effect were aware of which active agent had been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Treatment (Active Comparator): oral (250mg three times daily for 7 days) metronidazole
  Interventions: Drug: oral versus vaginal metronidazole
- Vaginal Treatment (Active Comparator): intravaginal (5 g of 0.75% gel twice daily for 5 days) metronidazole
  Interventions: Drug: oral versus vaginal metronidazole

INTERVENTIONS:
Drug: oral versus vaginal metronidazole

SUMMARY:
The goal of this study is to examine acceptability and efficacy of 2 kinds of BV treatment among women at low risk for preterm delivery. The objectives are:

1. To examine the side effects and patient acceptability of oral versus intravaginal metronidazole.
2. To compare the efficacy of oral and intravaginal metronidazole for the treatment of BV
3. To study the efficacy of oral and intravaginal metronidazole for the prevention of hospital admission during the 3rd trimester, chorioamnionitis, preterm delivery, and maternal infectious morbidity.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled intervention trial. Women diagnosed as BV+ by Gram stain at 12-16 weeks gestation are randomly assigned to the following treatment groups: oral metronidazole (250 mg TID x 7 days) with intravaginal placebo; intravaginal metronidazole (5g 0.75% gel BID x 5 days) with oral placebo. African American, Hispanic, Asian/Pacific Islander, Native American, and white women are eligible. Women with a prior preterm delivery, multiple gestation, chronic hypertension or pre-existing diabetes, antibiotic use before enrollment in the study, allergy to metronidazole, history of alcohol abuse in past year, and women under age 18 are excluded.

ELIGIBILITY:
Inclusion Criteria:

* Tested positive for bacerial vaginosis (Nugent score >7)
* African American, Hispanic, Asian/Pacific Islander, Native American, and white women

Exclusion Criteria:

* >20 weeks gestaion
* history of preterm delivery
* had a multiple gestation pregnancy
* had major medical complications (e.g., chronic hypertension or pre-existing diabetes)
* antibiotic use within 7 days of screening visit for enrollment in the study,
* allergy to metronidazole
* history of alcohol dependency in past year women under age 16

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 1999-10; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Microbiological, Clinical, and Therapeutic Cure Rates at Follow-Up among Women Treated with Oral vs. Intravaginal Metronidazole | 4 weeks after treatment
  Cure rates were assessed by Gram Stain Score (0-3, 4-6, 7-10); Abnormal clincial signs (0, 1-2, 3-4); Therapeutic cure (Gram Stain 0-3 and no symptoms) treatment

SECONDARY OUTCOMES:
preterm delivery | at delivery
  rate of delivery before 37 completed weeks gestation in intervention groups
low birth weight | at delivery
  birth weight less than 2500 grams

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Hitti, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell C, Balkus J, Agnew K, Lawler R, Hitti J. Changes in the vaginal microenvironment with metronidazole treatment for bacterial vaginosis in early pregnancy. J Womens Health (Larchmt). 2009 Nov;18(11):1817-24. doi: 10.1089/jwh.2009.1378. PMID 19951217
- [Background] Mitchell CM, Hitti JE, Agnew KJ, Fredricks DN. Comparison of oral and vaginal metronidazole for treatment of bacterial vaginosis in pregnancy: impact on fastidious bacteria. BMC Infect Dis. 2009 Jun 10;9:89. doi: 10.1186/1471-2334-9-89. PMID 19515236